CLINICAL TRIAL: NCT00253695
Title: Sleep Studies in HIV+ Older Children/Adolescents
Brief Title: Sleep, HIV Disease Progression, and Function in HIV Infected Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, William Shearer, Professor, Baylor College of Medicine
Other Study IDs: 1317; R01HL079533 (NIH)
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Sleep; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Wrist Actigraphy — Wrist actigraph will record participants' sleeping patterns.

SUMMARY:
This study is a first step in approaching the gap existing between understanding sleep abnormalities, alterations in sleep-regulating cytokines and HIV-1 disease regulating cytokines, and abnormal higher cortical function.

DETAILED DESCRIPTION:
BACKGROUND:

In the growing number of HIV infected youth and young adults, it is important to study the effects of HAART treatment on sleep patterns and related neurocognitive and psychosocial function.

DESIGN NARRATIVE (including primary and secondary outcomes):

Using validated sleep questionnaires and actigraphy measurements, overnight polysomnography (PSG, sleep study) will assess the degree of abnormal sleeping patterns and daytime sleepiness in HIV infected children and HIV uninfected children (control group).

The following peripheral blood levels will be measured over a 24-hour period, at multiple time points, in all participants: TNF-alphaRI and IL-6 (sleep-regulating cytokines); IFN-gamma and IL-12 (cytotoxic or TH1 cytokines); and IL-10 and IL-1RA (inflammatory or TH2 cytokines). This will help to determine the association between alterations in sleep-regulating cytokines and HIV disease progression (CD4+ T-cell count, HIV-1 RNA level).

Neurocognitive and neuropsychological tests will be performed on all participants to determine if there is an association between lack of normal sleeping habits, alterations in sleep-regulating cytokines and HIV-1 disease progression cytokines, and neurocognitive/neuropsychological performance.

Computer analysis of electroencephalography (EEG) will be performed during wakefulness and all stages of sleep to determine if greater disease severity, sleepiness, sleep disruption, and neurocognitive impairment is associated with increased amounts of slow activity. Improvement in these related factors will be associated with normalizations of these parameters. For some of these quantitative measures, the findings may be more significant for particular brain regions; for example, frontal regions in the case of attention problems.

ELIGIBILITY:
Inclusion Criteria:

HIV Group

* HIV-1 infection

Control Group

* Family members and friends of HIV-1 infected children

Exclusion Criteria:

HIV Group

* Pregnancy

Control Group

* Pregnancy
* Asthma
* Sleep apnea

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: HIV-infected children with and without asthma.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2004-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Association of cytokines, sleep patterns, and neurocognitive function in youth with HIV. | 11/2005 - 02/2009
  Observational study only

CONTACTS AND LOCATIONS:
Overall Officials: William Shearer, MD, PhD, Principal Investigator — Texas Children's Hospital/Baylor College of Medicine
Locations (1):
- Texas Children's Hospital/Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Foster SB, Paul ME, Kozinetz CA, Macias CG, Shearer WT. Prevalence of asthma in children and young adults with HIV infection. J Allergy Clin Immunol. 2007 Mar;119(3):750-2. doi: 10.1016/j.jaci.2007.01.002. No abstract available. PMID 17336620
- [Background] Foster SB, Paul ME, Glaze DG, Reuben JM, Harris LL, Cohen EN, Lee B-N, Kozinetz CA, Schwarzwald HL, Kline MW, Jackson CD, Loeb AJ, Frerking PR, Brouwers PY, Shearer WT. Viremia is associated with sleep disturbances, neurocognitive disorders and cytokine dysregulation in pediatric HIV infection. J Allergy Clin Immunol 2007;119;S232.
- [Background] Alvarez JA, Scully RE, Miller TL, Armstrong FD, Constine LS, Friedman DL, Lipshultz SE. Long-term effects of treatments for childhood cancers. Curr Opin Pediatr. 2007 Feb;19(1):23-31. doi: 10.1097/MOP.0b013e328013c89e. PMID 17224658
- [Background] Armstrong FD. Neurodevelopment and chronic illness: Mechanisms of disease and treatment. Ment Retard Dev Disabil Res Rev. 2006;12(3):168-73. doi: 10.1002/mrdd.20114. PMID 17061286
- [Background] Fisher SD, Miller TL, Lipshultz SE. Impact of HIV and highly active antiretroviral therapy on leukocyte adhesion molecules, arterial inflammation, dyslipidemia, and atherosclerosis. Atherosclerosis. 2006 Mar;185(1):1-11. doi: 10.1016/j.atherosclerosis.2005.09.025. Epub 2005 Nov 16. PMID 16297390
- [Background] Kozinetz CA, Matusa R, Hacker CS. Biologic and social determinants of sequelae and long-term survival of pediatric HIV in Romania. Ann Epidemiol. 2006 Aug;16(8):593-9. doi: 10.1016/j.annepidem.2005.11.012. Epub 2006 Jan 23. PMID 16431133
- [Background] Lewis DE, Gross KL, Diez MM, Martinez ML, Lukefahr HN, Kozinetz CA, Arduino RC. CD8 apoptosis may be a predictor of T cell number normalization after immune reconstitution in HIV. J Transl Med. 2007 Jan 30;5:9. doi: 10.1186/1479-5876-5-9. PMID 17263884
- [Background] Lipshultz SE, Fisher SD, Sharma T, Milton A, Miller TL. HIV-associated cardiovascular disease. Dialogues in Cardiology 2007, in press.
- [Background] Macias CG, Caviness AC, Sockrider M, Brooks E, Kronfol R, Bartholomew LK, Abramson S, Shearer W. The effect of acute and chronic asthma severity on pediatric emergency department utilization. Pediatrics. 2006 Apr;117(4 Pt 2):S86-95. doi: 10.1542/peds.2005-2000F. PMID 16777836
- [Background] Mitchell CD, Armstrong FD, Goodman KW, Cava A. Disclosure of HIV status to an infected child: medical, psychological, ethical, and legal perspectives in an era of "super-vertical" transmission. J Clin Ethics. 2008 Spring;19(1):43-52. No abstract available. PMID 18552052
- [Background] Nathan PC, Patel SK, Dilley K, Goldsby R, Harvey J, Jacobsen C, Kadan-Lottick N, McKinley K, Millham AK, Moore I, Okcu MF, Woodman CL, Brouwers P, Armstrong FD; Children's Oncology Group Long-term Follow-up Guidelines Task Force on Neurocognitive/Behavioral Complications After Childhood Cancer. Guidelines for identification of, advocacy for, and intervention in neurocognitive problems in survivors of childhood cancer: a report from the Children's Oncology Group. Arch Pediatr Adolesc Med. 2007 Aug;161(8):798-806. doi: 10.1001/archpedi.161.8.798. PMID 17679663
- [Background] Shearer WT, DeVille JG, Samson PM, Moye JH Jr, Fletcher CV, Church JA, Spiegel HM, Palumbo P, Fenton T, Smith ME, Graham B, Kraimer JM, Olson WC. Susceptibility of pediatric HIV-1 isolates to recombinant CD4-IgG2 (PRO 542) and humanized mAb to the chemokine receptor CCR5 (PRO 140). J Allergy Clin Immunol. 2006 Aug;118(2):518-21. doi: 10.1016/j.jaci.2006.03.028. Epub 2006 May 19. No abstract available. PMID 16890780
- [Background] Pacheco SE, McIntosh K, Lu M, Mofenson LM, Diaz C, Foca M, Frederick M, Handelsman E, Hayani K, Shearer WT; Women and Infants Transmission Study. Effect of perinatal antiretroviral drug exposure on hematologic values in HIV-uninfected children: An analysis of the women and infants transmission study. J Infect Dis. 2006 Oct 15;194(8):1089-97. doi: 10.1086/507645. Epub 2006 Sep 11. PMID 16991083
- [Background] Williamson MP, McCormick TG, Nance CL, Shearer WT. Epigallocatechin gallate, the main polyphenol in green tea, binds to the T-cell receptor, CD4: Potential for HIV-1 therapy. J Allergy Clin Immunol. 2006 Dec;118(6):1369-74. doi: 10.1016/j.jaci.2006.08.016. Epub 2006 Oct 13. PMID 17157668
- [Background] HIV Paediatric Prognostic Markers Collaborative Study. Predictive value of absolute CD4 cell count for disease progression in untreated HIV-1-infected children. AIDS. 2006 Jun 12;20(9):1289-94. doi: 10.1097/01.aids.0000232237.20792.68. PMID 16816558
- [Background] Fletcher CV, DeVille JG, Samson PM, Moye JH Jr, Church JA, Spiegel HM, Palumbo P, Fenton T, Smith ME, Graham B, Kraimer JM, Shearer WT; Pediatric AIDS Clinical Trials Group, Protocol 351 Study Group. Nonlinear pharmacokinetics of high-dose recombinant fusion protein CD4-IgG2 (PRO 542) observed in HIV-1-infected children. J Allergy Clin Immunol. 2007 Mar;119(3):747-50. doi: 10.1016/j.jaci.2006.10.045. No abstract available. PMID 17336619
- [Result] Foster SB, Lu M, Glaze DG, Reuben JM, Harris LL, Cohen EN, Lee BN, Zhao E, Paul ME, Schwarzwald H, McMullen-Jackson C, Clark C, Armstrong FD, Brouwers PY, Miller TL, Colin AA, Scott GB, Shahzeidi S, Willen EJ, Asthana D, Lipshultz SE, Thompson BW, Shearer WT. Associations of cytokines, sleep patterns, and neurocognitive function in youth with HIV infection. Clin Immunol. 2012 Jul;144(1):13-23. doi: 10.1016/j.clim.2012.04.004. Epub 2012 May 2. PMID 22659030